CLINICAL TRIAL: NCT02929472
Title: Effect of a Multicomponent Intervention on Physical Fitness and Metabolic Risk Markers in Children and Adolescents: A Pilot Study
Brief Title: Effect of a Multicomponent Intervention in Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clarice Maria de Lucena Martins (Other)
Responsible Party: Sponsor-Investigator, Clarice Maria de Lucena Martins, Professor PhD, Federal University of Paraíba
Organization: Federal University of Paraíba (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM-AF-RM
Record Dates: First submitted 2016-09-29; First posted 2016-10-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-09

CONDITIONS: Physical Activity; Metabolic Diseases
Keywords: Physical Activity; Physical Fitness; Intervention; Children and Adolescents
MeSH Terms: conditions — Motor Activity; Metabolic Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Exercise (Experimental): The intervention group (INT, n = 17, 7 boys) who attended at least 75% of PA classes and met more than 50% of food goals.The exercise sessions took 90 minutes, in order to assure at least 60 minutes of physical exercise, during 12 weeks. The sessions were always taught by the same staff, and were composed of: 10 minutes of warm-up; 30 minutes of circuit training; 15-minute of pre-sports and recreational games;and 5 minutes resting activities.
  Interventions: Behavioral: Physical exercise
- without physical exercise (Other): The control one (CONT, n = 18, 6 boys), with a minimum or less than 49% attendance in PA classes, and were not involved in the nutrition education program.
  Interventions: Behavioral: without physical exercise

INTERVENTIONS:
Behavioral: Physical exercise — The intervention group (INT, n = 17, 7 boys) who attended at least 75% of PA classes and met more than 50% of food goals.The exercise sessions took 90 minutes, in order to assure at least 60 minutes of physical exercise, during 12 weeks. The sessions were always taught by the same staff, and were composed of: 10 minutes of warm-up; 30 minutes of circuit training; 15-minute of pre-sports and recreational games;and 5 minutes resting activities.
  Arms: Physical Exercise
Behavioral: without physical exercise — The control one (CONT, n = 18, 6 boys), with a minimum or less than 49% attendance in PA classes, and were not involved in the nutrition education program.
  Arms: without physical exercise

SUMMARY:
The aim of this study was: to evaluate the effectiveness of a multicomponent pilot intervention in improving physical fitness (PF) and metabolic risk markers in children and adolescents; and examine if possible changes in PF are associated with metabolic risk markers in children and adolescents exposed to intervention. For such, a multicomponent pilot intervention was performed, consisting of sessions of physical exercise and nutrition education.The study included 35 children and adolescents (ages 7-13) divided into two groups: a intervention group (INT, n = 17) and a control one (CONT, n = 18). The sample underwent two moments of data collection (T0 and T1). The 1-hour exercise sessions were held based on an intensity above 65% of maximum HR. To assess the metabolic risk markers, analyzes of total cholesterol, HDL-C fraction, LDL-c fraction, triglycerides, blood glucose, insulin, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) were conducted in T0 and T1. Physical activity (PA) was assessed by accelerometry (Actigraph, GT3-X model, Florida) for 10 consecutive days. The health related PF components were evaluated throw different tests 20m Shuttle-run Test; handgrip dynamometry (TKK 5101 tightening D; Tokyo Japan); standing feet jump Test; Abdominal Test; trunk extension test; and body mass index (BMI) was calculated. Motor fitness was assessed by coordinations Test für Kinder - KTK. To assess food consumption, a 24-hour recall was held. For statistical analysis, the t-Student test and General Linear Model (GLM) - ANCOVA for repeated measures test with post-hoc Bonferroni (p <0.05) were performed. Multilinear regressions were done to analyse associations between measured outcomes.

DETAILED DESCRIPTION:
Study design

This quasi-experimental pilot study is part of a research study called "ACTION FOR HEALTH (Adolescents and Children in a Training InterventiON FOR HEALTH)", developed with youth of both gender (7-15 year-olds). It is a multicomponent intervention program to promote PA classes and nutrition education, and based on the behavior change Ecological Model. This information is hypothesis of the study.

ACTION FOR HEALTH study was approved by the Ethics Committee of the Center of Health Sciences of Federal University of Paraíba- Brazil (UFPB). The parents of the participants signed out a consent term.

Study sample The project was announced in public and private schools of João Pessoa (Brazil), as well as through print (newspapers) and electronic (social network) media. 59 youth volunteered, and 43 children and adolescents (7-13 year-olds) met the eligibility criteria. 8 of them did not complete all the study protocol.

So, 35 comprised the sample and did all the evaluation protocol. Participants were divided in two groups: the intervention group (INT, n = 17, 7 boys) who attended at least 75% of PA classes and met more than 50% of food goals; and the control one (CONT, n = 18, 6 boys), with a minimum or less than 49% attendance in PA classes, and were not involved in the nutrition education program.

Methodologies study and preparation of the intervention The program was developed by 4 teachers, 7 graduate students, 1 nutritionist, 2 graduate Nutrition students, and 1 cardiologist, and participated in weekly meetings where methodologies and intervention sessions were prepared and tested. During this test period, activities that would promote greater adherence of students were listed. Additionally, participants randomly used a heart rate monitor (Polar Team2 Pro, Polar, Finland) and an accelerometer (Actigraph, GT3X model), in order to record activities that promoted more significant increases in heart rate and in moderate and vigorous PA intensities.

Physical exercise intervention The exercise sessions took 90 minutes, in order to assure at least 60 minutes of physical exercise, during 12 weeks. The sessions were always taught by the same staff, and were composed of: 10 minutes of warm-up; 30 minutes of circuit training; 15-minute of pre-sports and recreational games;and 5 minutes resting activities.

Warm-up included aerobic/anaerobic and recreational activities. The circuit, divided into 6 stations, included activities that prioritized conditional and/or coordinative physical capacities, accordingly with the purpose of the proposed session for the day, so that participants could maintain a high intensity throughout the circuit.

In the first month, the duration of each circuit station was 30 seconds, which was increased to 45 seconds and 60 seconds, in the second and third month, respectively. The transition time between each station was kept in 30 seconds throughout the intervention. Finally, low-heart rate activities were carried out, with games to music and stretching.

The intensity of the training sessions was defined in a heart rate (HR) average over 65% of maximum heart rate of each participant.

Nutritional education intervention The dietary intervention, designed by the nutritionist staff, consisted of two actions. The first was trough monthly events throughout the intervention, one in the beginning of each month, with participation of participants' parents. The second action consisted on the achievement of 3 dietary goals (an easy, an average and hard goal) to which children and adolescents should meet during the months of intervention. These goals were added during the intervention, so that the beginning of the 1st month of intervention participants had three goals to meet, and at the beginning of the 3rd month, 9 goals. They also received a worksheet to record if they met the minimum (1 star), average (2 stars) and maximum (3 stars) of the daily goal.

Parental support Simultaneously, exercise sessions were offered to parents in order to encourage family participation in the intervention performed with children and adolescents. The activities were carried out by a volunteer PA teacher in the center of sports of UFPB.

Study variables Sexual maturation Each participant self-assessed their own stage of secondary sexual characteristics: breast development stage in women and pubic hair in males (TANNER, 1962). The correlation between self-assessment of sexual maturity state and evaluation performed by the parent was 78% for female and 90% male. This variable was used as confounder in the statistical procedures.

Anthropometric measure Height, determined by a stadiometer "Holtain", followed the standard procedure of Lohman (1988). Two measurements were performed, recorded in meters to the nearest millimeter, and was considered the arithmetic mean of the two measurements. Body composition was measured after 4-hour-fasting and low water intake, and then, a bioimpedance scale was used (Inbody 720, Biospace Co., Ltd.) to determine body weight and fat mass.

Metabolic variables Blood samples from the participants were collected after a nocturnal 12 hour-fasting, by laboratory specialists, through peripheral puncture in the cubital vein. The analysis of CT, HDL-C, triglyceride, and glucose was carried out by spectrophotometry (Cobas Integra 400 Plus) with Roche® kits. The LDL-C fraction was indirectly calculated using the Friedewald formula (1972). The aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels were determined by enzyme kinetic assay for spectrophotometrically obtained after centrifugation 10 minutes / 3500 rpm. Insulin was determined by Luminex-100 IS (Integrated System: Luminex Corporation, Austin, TX, USA), using the Linco Human Gut Hormone panel kit (Linco Research Inc., MO, USA). The insulin resistance was determined by HOMA-IR.

Physical activity and sedentary behavior PA was measured by accelerometer (Actigraph, GT3X model, Florida). The participants used an accelerometer for 10 consecutive days, and they also received instructions for the correct use of the device. At the time of explanation and visual demonstration of the proper use of the device, participants received a list of instructions, along with a diary of activities in which they were required to record wear and non-wear time of the instrument, and also habitual physical activities.

Data reduction was performed by Actlife software, version 6.11.7. For the validation data, at least 4 days of recording at least 8 hours per day (480 minutes / day) were considered 40. Of these 4 days, 2 days corresponded to the intervention and 2 without intervention (1 weekend day). The time of non-use was estimated based on periods of more than 20 consecutive minutes of zero. For data download, 15 seconds epochs were performed, based on recommendations to similar populations. The useful and non-time has been determined according to Troiano (2007). The cutoff points for determining the time spent on different intensities of PA followed the standards proposed by Evenson et al (2008). To determine time spent for physical activity /week in each of the intensities was necessary to perform a calculation to generate weighted averages in minutes / day, of PA intensities. Time spent in moderate-to-vigorous physical activity corresponded to the sum of moderate physical activity (AFM) and vigorous physical activity (AFV) values.

Health related Physical Fitness Health related Physical Fitness components were evaluated from different tests of Fitnessgram battery test (1999) and ALPHA battery test, which those protocols were performed internationally for similar populations. Thus, cardiorespiratory fitness (CRF) was measured using the test-run Suttle 20 m. The test was complete when the participant failed to reach the final lines simultaneously with the audio signals on two consecutive occasions, or when it ended the test due to fatigue.

Muscle strength of upper limbs was measured by handgrip dynamometer with adjustable pinch (TKK 5101 Grip D; Takey, Tokyo Japan), which was conducted twice on each hand and recorded the maximum score achieved in kilograms. For analysis, it was calculated a mean value between the measurements of each hand. Muscle strength of the lower limbs was assessed by Jumping test with feet together. The participant leaped forward as much as possible, on a stable, non-slip surface. The test was performed twice and the best score was recorded in centimeters. Abdominal strength and endurance were measured by repetitions of abdominal test, when the participant had to perform a maximum possible number of sit-ups, up to a maximum of 75 for one minute.

Trunk strength and flexibility were assessed by trunk extension test. There were performed two attempts and validated the best one. Flexibility of the lower limbs was assessed by sit-and-reach test, and were performed two attempts for each leg and used the average value between the two attempts for each leg. Body composition was measured by body mass index (BMI), calculated using the formula (weight / height) 2. Motor fitness was evaluated by Koordinations Test für Kinder Tests - KTK battery of tests, which is recommended for evaluation of motor components such as balance, coordination, speed and agility, in children.

Food consumption Food consumption was carried out by a 24-hour recall. Participants, along with their parents informed food consumption during the past two weekdays and one weekend day before evaluation. Data from the three days were tabulated in the software "Virtual Nutri", to calculate the total energy consumption values for each of the three days. For analytical procedures, it calculated the average caloric intake among the three measurements.

ELIGIBILITY:
Inclusion Criteria:

* volunteered to participate in the study
* Excess weight / obesity for experimental group
* Aged 7 to 13 years

Exclusion Criteria:

* No complete evaluation protocol

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2015-05; Primary Completion 2015-06 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
cardiorespiratory fitness | 3-months
  Shuttle-run Test 20m - participants ran between two lines 20m away, keeping the rhythm corresponding to the audio signals from a prerecorded CD. The initial speed was 8.5km / h and increased 0.5km / h every minute (one minute corresponds to one stage). Participants were instructed to run in a straight line, at their own pace, and returning at the end of each beep. The test was completed when the participant failed to reach the final lines simultaneously with the audio signals on two consecutive occasions, or when it ended the test due to fatigue. The procedure was done previously described by Leger et al (1988).
Muscle strength of the upper limbs | 3-months
  Pinch manual - using a manual dynamometer with adjustable pinch (TKK 5101 Grip D; Takey, Tokyo Japan). The participant held a gradual and continuous hold for at least two seconds, with the right and left hand, with the elbow in full extension as standard procedure described above (CENTERS FOR DISEASE CONTROL AND PREVENTION (CDC). NATIONAL CENTER FOR HEALTH STATISTICS ( NCHS), 2011). The test was conducted twice on each hand and recorded the maximum score achieved in kilograms. For analysis it computed the average value between the measurements of each hand.
muscle strength of the lower limbs: | 3-months
  jump test with feet together - from an initial position with your feet parallel, immediately behind a line drawn on the ground, the participant leaped forward as much as possible, on a hard, non-slip surface. The test was performed twice and the best score was recorded in centimeters.
Abdominal endurance: | 3-months
  Test repetitions of abdominal - was to make the largest possible number of sit-ups, up to a maximum of 75 for one minute. Lying on a mattress with your knees bent, arms straight, palms face down and his head resting on the mattress. a banner was placed with a width of 11.5 cm, under the performer's knees. This track was used to determine the route to be traveled by sliding your hands on the mattress.
Flexibility of the trunk: | 3-months
  trunk extension test - consisted of starting from the prone position, with legs and outstretched arms and hands under the thighs, raise trunk controllably up to a maximum of 30 cm (measured between your chin and the mattress). There were two attempts and validated the best of them.
Flexibility of the lower limbs: | 3-months
  Test sit and reach - was to achieve the greatest distance possible with your hands, one over the other, with the participant barefoot, with the left leg bent and the other with the foot flat on the measuring bench. There were two attempts for each leg and used the average value between the two attempts for each leg.
Body composition: | 3-months
  body mass index (BMI) - was calculated using the formula (weight / height) 2.

SECONDARY OUTCOMES:
Cholesterol Markers | 3-months
  Blood samples from the participants were collected after a nocturnal 12 hour-fasting, by laboratory specialists, through peripheral puncture in the cubital vein. The analysis of CT, HDL-C was carried out by spectrophotometry (Cobas Integra 400 Plus) with Roche® kits. The LDL-C fraction was indirectly calculated using the Friedewald formula (1972).
Hepatic markers | 3-months
  Blood samples from the participants were collected after a nocturnal 12 hour-fasting, by laboratory specialists, through peripheral puncture in the cubital vein.The aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels were determined by enzyme kinetic assay for spectrophotometrically obtained after centrifugation 10 minutes / 3500 rpm.
Insulin | 3-months
  Blood samples from the participants were collected after a nocturnal 12 hour-fasting, by laboratory specialists, through peripheral puncture in the cubital vein. Insulin was determined by Luminex-100 IS (Integrated System: Luminex Corporation, Austin, TX, USA), using the Linco Human Gut Hormone panel kit (Linco Research Inc., MO, USA). The insulin resistance was determined by HOMA-IR
Triglycerides | 3-months
  Blood samples from the participants were collected after a nocturnal 12 hour-fasting, by laboratory specialists, through peripheral puncture in the cubital vein. The analysis of TGL, was carried out by spectrophotometry (Cobas Integra 400 Plus) with Roche® kits.
Glucose | 3-months
  Blood samples from the participants were collected after a nocturnal 12 hour-fasting, by laboratory specialists, through peripheral puncture in the cubital vein. The analysis of glucose was carried out by spectrophotometry (Cobas Integra 400 Plus) with Roche® kits.

IPD SHARING:
Plan to Share IPD: No